CLINICAL TRIAL: NCT01027494
Title: Topical Treatment of Acute Otitis Media Through Tympanostomy Tubes (AOMT) and Its Effect on Microbial Flora Distal to the Site of Infection
Brief Title: Topical Treatment of Acute Otitis Media Through Tympanostomy Tubes (AOMT) and Its Effect on Microbial Flora
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: C-09-017
Record Dates: First submitted 2009-12-04; First posted 2009-12-08 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Acute Otitis Media
Keywords: ear tubes; ear drainage; ear infection; ear drops; tympanostomy tubes
MeSH Terms: conditions — Otitis Media; Otitis | interventions — Ciprofloxacin; Dexamethasone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment: Ciprofloxacin 0.3% and dexamethasone 0.1% otic suspension, 4 drops in outer ear canal of infected ear(s) while awake 2 times per day for 7 days
  Interventions: Drug: Ciprofloxacin 0.3% and dexamethasone 0.1% otic suspension
- Healthy: No intervention

INTERVENTIONS:
Drug: Ciprofloxacin 0.3% and dexamethasone 0.1% otic suspension — Four drops in the outer ear canal of infected ear(s) while awake 2 times per day for 7 days
  Other Names: CIPRODEX®
  Groups: Treatment

SUMMARY:
The purpose of this observational study was to evaluate the effects of a topical fluoroquinolone (antibiotic) instilled into the otic (ear) canal to treat Acute Otitis Media through Tympanostomy Tubes (AOMT) on selected bacterial species on the skin near the ear, in the nose, and in the throat.

DETAILED DESCRIPTION:
Pediatric patients with tympanostomy tubes were enrolled into one of two groups: 1) Treatment, i.e., patients with signs of otic infection, to be treated with CIPRODEX; or 2) Healthy, i.e., patients without signs of otic infection, to receive no treatment. Microbiological specimens were collected from four areas (ear canal, skin, nose, throat) during three study visits (Day 1, Day 8, and Day 42), and the specimens collected from the Healthy group served as a comparison (control) group for identifying fluoroquinolone (FQ) resistant bacterial strains.

ELIGIBILITY:
Inclusion Criteria:

* Six months to less than 5 years of age at time of enrollment;
* Presence of bilateral, patent tympanostomy tubes;
* Otorrhea-free for at least 7 days following tympanostomy tube surgery (healthy group);
* Otorrhea up to and including 21 days in duration in at least one ear at Visit 1 (treatment group);
* Willing to refrain from significant water immersion of both ears without the use of adequate ear protection during swimming, bathing, showering and other water-related activities;
* Read and sign informed consent (parent or guardian);
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Ongoing/current therapy as described in protocol;
* Has received any treatment for current AOMT episode (treatment group);
* Otorrhea greater than 21 days in duration immediately prior to Day 1 visit (treatment group);
* History of or current acute or chronic non-tube otorrhea (through existing perforation of the eardrum);
* Current acute otitis externa (AOE), or malignant otitis externa (MOE) or other conditions which could interfere with evaluation of the study drug;
* Known or suspected ear infection of fungal or mycobacterial origin (treatment group);
* History or active herpes simplex, vaccina or varicella infections or overt viral infection of the tympanic membrane or the external canal;
* Prior otologic surgery, except that confined to the tympanic membrane, within one year of study entry;
* Diabetes;
* Any current known or suspected infection (other than AOMT) requiring systemic antimicrobial therapy;
* Known or suspected allergy or hypersensitivity to quinolones;
* Other protocol-defined exclusion criteria may apply.

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants were selected from medical practices serving pediatric patients.
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2009-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in microbial organism susceptibility and fluoroquinolone resistant flora at sites distal to the original infection. | 42 + 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Gale Cupp, MS, Study Director — Alcon Research
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States